CLINICAL TRIAL: NCT00228345
Title: The Significance of Glucose Intolerance in the Pathogenesis of Idiopathic Axonal Polyneuropathy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study Completed
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12896A
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Idiopathic Axonal Polyneuropathy; Abnormal OGTT
Keywords: Idiopathic Axonal Polyneuropathy; abnormal OGTT
MeSH Terms: interventions — Tomography, Optical Coherence

INTERVENTIONS:
Procedure: Optical coherence tomography,Fluorescein angiography

SUMMARY:
The purpose of this study is to determine whether impaired glucose handling (abnormality in the way the body processes blood sugar) can cause a neuropathy (damage to the nerves).

DETAILED DESCRIPTION:
Neuropathy of undetermined etiology is a common disease that usually starts at the sixth to seventh decades. It can cause significant pain and disability. Previous studies have demonstrated increased prevalence of abnormal glucose handling, when these patients were tested with oral glucose tolerance test (OGTT). On the other hand, many of the neuropathy patients suffer from pain and depression and obesity; and abnormal OGTT in these patients may be the result of these factors. We assume that if abnormal handling of blood sugar is the cause of neuropathy, these patients may have evidence of damage to other organs (like eyes and kidneys) as a result of abnormal blood sugar. In a pilot study, we will determine the incidence of subtle damage to kidneys, eyes and also look for other factors associated with abnormal glucose handling in patients with neuropathy and abnormal OGTT and compare it to age matched controls with normal OGTT.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria (for the subjects) will include peripheral neuropathy, age more than 50 years, and a negative workup for neuropathy (aside from an abnormal OGTT). Age matched controls will have no history of diabetes or baseline retinal disease . A workup to rule out other causes of peripheral neuropathy, and an OGTT, will be performed prior to participation in the study.

Exclusion Criteria:

Patients with abnormal OGTT in the diabetic range will not be included.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-01; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
we will determine the incidence of subtle damage to kidneys, eyes and also look for other factors associated with abnormal glucose handling in patients with neuropathy and abnormal OGTT and compare it to age matched controls with normal OGTT. | 48 hrs

SECONDARY OUTCOMES:
we will determine the incidence of subtle damage to kidneys, eyes and also look for other factors associated with abnormal glucose handling in patients with neuropathy and abnormal OGTT and compare it to age matched controls with normal OGTT | 48 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Kourosh Rezania, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Dive D, Lievens I, Moonen G, Wang FC. [Diabetic peripheral neuropathy]. Rev Med Liege. 2005 May-Jun;60(5-6):490-7. French. PMID 16035316
- [Background] 1. McLeod, J.G., et al., Chronic polyneuropathy of undetermined cause. J Neurol Neurosurg Psychiatry, 1984. 47(5): p. 530-5. 2. Dyck, P.J., K.F. Oviatt, and E.H. Lambert, Intensive evaluation of referred unclassified neuropathies yields improved diagnosis. Ann Neurol, 1981. 10(3): p. 222-6. 3. Wolfe, G.I., et al., Chronic cryptogenic sensory polyneuropathy: clinical and laboratory characteristics. Arch Neurol, 1999. 56(5): p. 540-7. 4. Notermans, N.C., et al., Chronic idiopathic polyneuropathy presenting in middle or old age: a clinical and electrophysiological study of 75 patients. J Neurol Neurosurg Psychiatry, 1993. 56(10): p. 1066-71. 5. Beghi, E. and M.L. Monticelli, Chronic symmetric symptomatic polyneuropathy in the elderly: a field screening investigation of risk factors for polyneuropathy in two Italian communities. Italian General Practitioner Study Group (IGPST). J Clin Epidemiol, 1998. 51(8): p. 697-702. 6. Notermans, N.C. and J.H. Wokke, Chronic idiopathic axonal polyneuropathy. Muscle Nerve, 1996. 19(12): p. 1637-8. 7. Dyck, P.J., Cryptogenic sensory polyneuropathy. Arch Neurol, 1999. 56(5): p. 519-20. 8. Wolfe, G.I. and R.J. Barohn, Cryptogenic sensory and sensorimotor polyneuropathies. Semin Neurol, 1998. 18(1): p. 105-11. 9. Monticelli, M.L. and E. Beghi, Chronic symmetric polyneuropathy in the elderly. A field screening investigation in two regions of Italy: background and methods of assessment. The Italian General Practitioner Study Group (IGPSG). Neuroepidemiology, 1993. 12(2): p. 96-105. 10. Beghi, E. and M.L. Monticelli, Diabetic polyneuropathy in the elderly. Prevalence and risk factors in two geographic areas of Italy. Italian General Practitioner Study Group (IGPSG). Acta Neurol Scand, 1997. 96(4): p. 223-8.